CLINICAL TRIAL: NCT03147456
Title: Protein Supplementation Impact On Body Muscle Mass And Fat Mass In Qataris Post Bariatric Surgery, Randomized Controlled Trials (Rcts)
Brief Title: Protein Supplementation Impact On Body Muscle Mass And Fat Mass In Qataris Post Bariatric Surgery, Randomized Controlled Trials (Rct)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 16433
Record Dates: First submitted 2017-04-18; First posted 2017-05-10 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-03

CONDITIONS: Obesity
Keywords: bariatric; obesity; protein supplements
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Investigators and researchers in this study will be blinded to the intervention, i.e. they will not be aware of who is on protein supplement and who is on placebo. Patients will also be blinded to the intervention, i.e. they will not know whether they are taking protein or zero protein supplement. For the blinding there will be a dietician who will assign the treatment and the control to patients as per the above randomization results. This dietician will also be responsible for filling the intervention & control ready-to-feed shakes into identical bottles labeled either A or B, the dietician will not have any other responsibility such as data entry or follow up of participants as this will be done by the PI and research team, he will only be responsible for the blinding process.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients will receive nutritional counseling by a bariatric dietitian in a routine round, aiming that they will know the post-surgery diet stages and to not develop any nutritional deficiencies.Before discharge from the hospital, patients will receive supplement and will be advised by the dietitian regarding its use (one can per day, over 3-5 intervals). Supplement contains (per 200 ml can) 20 g of protein, 250Kacl plus different micronutrient and macronutrient (Cubitan Protein, Nutricia, Netherlands).
  Interventions: Dietary Supplement: (Cubitan Protein, Nutricia, Netherlands).
- Control group (Placebo Comparator): Patients will receive nutritional counseling by a bariatric dietitian in a routine round, aiming that they will know the post-surgery diet stages and to not develop any nutritional deficiencies. Before discharge from the hospital, patients will receive supplement and will be advised by the dietitian regarding its use (one can per day over 3-5 intervals).Following hospital discharge, Control patients will receive supplement contains per can (200 ml), 0g protein, fat free, 100 kcal and enriched with electrolytes (preOp, Nutricia, Netherlands).
  Interventions: Dietary Supplement: (preOp, Nutricia, Netherlands).

INTERVENTIONS:
Dietary Supplement: (Cubitan Protein, Nutricia, Netherlands). — Supplement contains (per 200 ml can) 20 g of protein, 250Kacl plus different micronutrient and macronutrient.
  Arms: Intervention group
Dietary Supplement: (preOp, Nutricia, Netherlands). — contains per can (200 ml), 0g protein, fat free, 100 kcal and enriched with electrolytes
  Arms: Control group

SUMMARY:
One of the most common post-operative deficiencies or complications of bariatric surgery is protein malnutrition. It may lead to many predicaments such as malnutrition, vitamin, micro- and macronutrient deficiencies that can lead to deleterious consequences. A protein-rich diet make a person feel satiety and thereby the consumption will be low in overall energy intake. The objectives of our study are. The aim of this study is to assess the effect of protein supplementation on changes in health parameters such as fat mass, muscle mass, weigh change, protein (total and albumin), Vit B12, Zinc and Magnesium, in Qatari patients post bariatric surgery. Our participants are Qatari aged 18-45 years males and females recruited from the bariatric surgery centers of 2 major HMC hospitals (HGH hospital) and will be randomized to receive either the protein supplement (treatment group) or a dietary advice (control group). All participants will be equally followed and monitored for 3 months and data on the above parameters will be collected, together with other population characteristics, at Baseline, 1 month and 3 month. Data will then be analyzed using the most up-to-date SPSS statistical package to assess the effect of protein supplementation on the parameters of interest. Statistical measures will be carefully chosen to properly assess the difference in the treatment (protein supplementation) effect compared with the control (Dietary advice). Investigators hypothesize that Patients receiving protein supplement (intervention group) Compared with patient not on protein supplement (placebo group) will maintain weight loss and other essential health parameters.

ELIGIBILITY:
Inclusion Criteria:

Study participants must have the following criteria in order to participate in the trial:

1. Qatari males or females.
2. Aged between 18 and 60 year
3. Based at the bariatric surgery list of HMC with their follow up scheduled be at HMC.

Exclusion Criteria:

Patients will be excluded from participating in the trial if they have the following criteria:

1. Any Renal or liver disease because that will affect protein or albumin level in body.
2. Past history of bariatric surgery
3. Patients will be further excluded after starting the trial if they fall into the following categories:

   * Subjects who did not take at least 80% of their intervention product amount per day, or
   * Subjects who did not comply with the treatment (or placebo) for more than 3 days per week.

Also, patients who refuse to participate & patients with baseline tests showing they are in need for protein supplements will be excluded from the study and given the needed protein supplements per the standard care.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-03-08 (Actual); Primary Completion 2017-08-01 (Estimated); Study Completion 2017-08-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of changes in Body Weight | 3 months
  Measurement of changes in Body Weight
Measurement of changes in Muscle mass. | 3 months
  Measurement of changes in Muscle mass.
Measurement of changes in Fat mass. | 3 months
  Measurement of changes in Muscle mass.

SECONDARY OUTCOMES:
To assess the measurement on Protein | 3 months
  To assess the measurement on Protein
To assess the measurement on Vitamin B12 | 3 months
  To assess the measurement on Vitamin B12
To assess the measurement on Magnesium | 3 months
  To assess the measurement on Magnesium
To assess the Zinc level measurement | 3 months
  To assess the Zinc level measurement

CONTACTS AND LOCATIONS:
Locations (1):
- sahar Dahawi Alshamari, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al-Shamari SD, ElSherif MA, Hamid W, Hanna F. The effect of protein supplementation on body muscle mass and fat mass in post-bariatric surgery: a randomized controlled trial (RCT) study protocol. Arch Public Health. 2018 Jan 22;76:7. doi: 10.1186/s13690-017-0252-2. eCollection 2018. PMID 29423219